CLINICAL TRIAL: NCT04021836
Title: Three Dimensional Evaluation of Nasolabial Changes Following Classic vs Without Alar Base Suture After Le Fort I Osteotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Afraa Bushra Abdelkarim Jubara, Dr afraa bushra abdelkarim jubara, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3DENB
Record Dates: First submitted 2019-07-13; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Quality of Life

STUDY DESIGN:
Intervention Model Description: Three dimensional evaluation of nasolabial changes following classic vs without alar base suture after Le Fort I osteotomy
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3d evaluation of naso labial changes using alar cinch suture (Other)
  Interventions: Other: 3d evaluation of nasolabial change
- 3d evaluation of nasolabial change without Alar cinch (Other)
  Interventions: Other: 3d evaluation of nasolabial change

INTERVENTIONS:
Other: 3d evaluation of nasolabial change — Evaluation of With vs without ala cinch suture after lefort 1 osteotomy

SUMMARY:
Three dimensional evaluation of nasolabial changes following classic vs without alar base suture after

Le Fort I osteotomy

A randomized controlled clinical trial

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with skeletal maxillomandibular deformity indicated for surgical correction by Le Fort I osteotomy.
2. Absence of growth.
3. Patients must be willing for the surgical procedure and follow-up, with his informed consent.

Exclusion Criteria:

* 4. History of facial trauma with fractures of facial bones. 5. History of surgical operation in nasal region. 6. Facial asymmetry. 7. Patients with accompanying craniofacial syndromes. 8. Patients with any diseases that compromise bone or soft tissue healing. 9. Anterior open bite cases. 10. Clefts ( lip and palate). 11. Medically compromised patients not fit for general anaesthesia. 12. missing preoperative or postop-erative 3D photographs or CBCT scans 13. multi-segment Le Fort I osteotomy 14. rhinoplasty surgery during or within 1 year after the Le Fort I osteotomy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
Widening of alar base | 6 months
  Widening of alar base

SECONDARY OUTCOMES:
Nasal volume | 6 months
  Nasal volume

IPD SHARING:
Plan to Share IPD: Yes